CLINICAL TRIAL: NCT06014749
Title: Analgesic Efficacy of Serratus Intercostal Block Versus Epidural Analgesia in Eventration Surgery : Prospective Observational Study
Brief Title: Serratus Intercostal Block Versus Epidural Analgesia in Eventration: Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Judith Andres, MD, Hospital del Rio Hortega
Other Study IDs: 22-EO132
Record Dates: First submitted 2023-08-02; First posted 2023-08-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Eventration; Regional Anesthesia; Epidural; Anesthesia; Abdominal Hernia
Keywords: Intercostal nerves, epidural,abdominal hernia
MeSH Terms: conditions — Gastroschisis; Hernia, Abdominal | interventions — Ultrasonography; Anesthesia, Conduction; Anesthetics, Local

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patient under serratus intercostal plane block: patients who will undergo a modified bilateral ultrasound-guided BRILMA block (SIPB) using a high-frequency linear probe (6-15 Hz) and 80 mm needle.
  Interventions: Procedure: undergo; Device: ultrasound; Drug: Local anesthetic
- patient under epidural analgesia: patients who undergo Epidural Analgesia prior to General Anesthesia and fentanyl 1 mcg/kg approx according to characteristics and needs and upon arrival at the URPA is connected to the PC Levobupi 0.125% at 6 ml / h + rescue boluses of Levobupi 0.125% 4 ml if needed in the 1st hours.
  Interventions: Procedure: undergo; Device: ultrasound; Drug: Local anesthetic

INTERVENTIONS:
Procedure: undergo — regional anesthesia
  Other Names: Eventroplasty
Device: ultrasound — ultrasound guided
  Other Names: Regional anesthesia
Drug: Local anesthetic — local anesthetic
  Other Names: Regional anesthesia

SUMMARY:
Adequate pain control, rehabilitation and early postoperative recovery are currently the model to follow according to the recommended guidelines.In this project the main objective is to evaluate 2 different analgesic strategies both intraoperatively and postoperatively, one based on 1. Epidural analgesia and the other 2. Echoguided serratus intercostal block prior to surgical intervention in eventration or abdominal wall repair interventions.

We conducted an observational study with a low level of intervention. Epidural analgesia prior to general anesthesia and serratus-intercostal block prior to general anesthesia) following the criteria applied in each case according to the operating room anesthesiologist until reaching the sample size and fulfilling the criteria of: abdominal eventration repair, over 18 years of age, ASA I-III. Signature of the IC.

DETAILED DESCRIPTION:
Adequate pain control, rehabilitation and early postoperative recovery are currently model to follow according to the recommended guidelines.In this project the main objective is to evaluate 2 different analgesic strategies both intraoperatively and postoperatively, one based on 1. Epidural analgesia and the other 2. Echoguided serratus intercostal block prior to surgical intervention in eventration or abdominal wall repair interventions.

The investigators conducted an observational study with a low level of intervention. Epidural analgesia prior to general anesthesia and serratus-intercostal block prior to general anesthesia) following the criteria applied in each case according to the operating room anesthesiologist until reaching the sample size and fulfilling the criteria of: abdominal eventration repair, over 18 years of age, ASA I-III. Signature of the IC.

We will assess the analgesia provided by both techniques and to compare the results.

ELIGIBILITY:
Inclusion Criteria:

* abdominal eventration repair,
* over 18 years old,
* ASA I-III.
* Signature of the IC.

Exclusion Criteria:

* Allergy to Local anesthetic

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people undergoing to repair abdominal wall
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain management | 24h
  Pain control. NRS scale at O,6, 12 and 24 h in postoperative time
postoperative quality of recovery | 24h
  Quality of recovery, QoR15 scale, that includes physical and psicological item. That scale will be fill by the patient 24 h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: María T Fernandez, MD, Study Director — Hospital del Rio Hortega
Locations (1):
- Judith Andres, Valladolid, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: Undecided
During the first year the preliminary results will be ready and will be present as abstract. Th estimated time to finish the study is 2 years